CLINICAL TRIAL: NCT03459976
Title: HE4 is a Beneficial Biomarker in Endometrial Cancer
Acronym: HE4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, f m dabnon, dr.fatma mohamed dapnon abuktaa, Ain Shams University
Other Study IDs: HE4 in endometrial cancer
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2 groups: control group case group
  Interventions: Diagnostic Test: evaluate serum level HE4 in endometrial cancer

INTERVENTIONS:
Diagnostic Test: evaluate serum level HE4 in endometrial cancer — 1. HE4 in beignin endometrial diseases
  2. HE4 in endometrial cancer

SUMMARY:
Evaluation of Serum level of Human Epididymis Secretory Protein 4 (HE4) in Endometrial Cancer and clinical significant it

DETAILED DESCRIPTION:
.Endometrial cancer represents the most common gynecologic cancer, and it is expected to become an even greater public health concer as the prevalence of obesity, one of the most common risk factors for endometrial cancer, increases worldwide, Approximately 42,160 cases are diagnosed annually, 7,780 deaths occur, and more than 4,000 new cases are diagnosed yearly (Renehan et al., 2008).

National Cancer Institute (NCI) statistics shows that while there was an. insignificant decline in the incidence of endometrial cancer (EC) from 1997 to 2006 (-0.4 annual percentage change), the mortality rate increased significantly in the same time period (+0,3 annual percentage change). These data seem to suggest a trend for an increasing frequency of more aggressive forms of EC in the United States, which underscores the need for a better understanding of the molecular mechanisms and pathways involved in EC pathogenesis (National Cancer Institute, 2013).

The diagnosis is usually done at an early stage, and approximately 70% of endometrial cancers are diagnosed as stage I; this results in better prognosis, with a 5-year overall survival rate of 90% to 95% (Jemal et al., 2009).

Almost 20% of patients with endometrial cancer are in the premenopausal state and 10% are asymptomatic. In such a case, it is much harder to make an early diagnosis and usually they are probably diagnosed at advanced stages (Li et al., 2009).

An earlier diagnosis represents an imperative goal to improve survival and prognosis of patients of endometrial cancer. Actually, there are no certified screening tools for endometrial cancer. Pelvic ultrasound as screening for endometrial cancer reaches 80.5% of sensitivity, when endometrial echo is > 5 mm, but it dramatically decreases to 20% in asymptomatic women; moreover, specificity is low (61%) (Jacobs et al., 2011).

HE4, a putative protease inhibition containing two (Whey Acid Protein) WAP domains, is significantly increased in the endometrioid subtype of EC (Drapkin et al., 2005).

Tissue microarray and real-time ploymerais chain reaction PCR studies confirmed a high level of HE4 expression in both endometrioid and serous types of EC (Jiang et al., 2013), these results are consistent with those from other laboratories showing increased HE4 mRNA and protein expression in endometrial cancer tissues (Moore el al., 2008; Bignotti et al., 2011).

Subsequent investigation demonstrated that HE4 are detectable in various normal tissues with varying expression levels, yet their levels are significantly increased in EC compared to normal endometrium (Jiang et al., 2013).

ELIGIBILITY:
Inclusion Criteria:

Age (40 - 70 yr old).

Exclusion Criteria:

1. Age more than 70 yr and less than 40 yr.
2. Abnormal cardiac hematological renal hepatic functions.
3. Breast cancer or other malignancies.
4. Concomitant benign and for malignant adnexal pathologies.
5. Hormonal medication.
6. Patient taking or having chemo-radiotherapy.
7. Patients unfit for surgical intervention.
8. Smoker.

Ages: 40 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Control group: 40 Patients with abnormal vaginal bleeding and diagnosed benign endometrial pathology by endometrial biopsy.
  Case group: 45 Patients with abnormal vaginal bleeding and diagnosed endometrial cancer at prior endometrial biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
: Evaluation of Serum Level of(HE4) in Benign Endometrial disease and Endometrial Cancer | 1 yeare
  * Evaluation of Serum Human Epididymis Secretory Protein 4 (HE4) in Benign Endometrial Endometrial Cancer Disease and
  * Evaluation of Serum Human Epididymis Secretory Protein 4 (HE4) in Benign Endometrial Endometrial Cancer Disease and
    c: Evaluation of Serum Human Epididymis Secretory Protein 4 (HE4) in Benign Endometrial Endometrial Cancer Disease and cas cotrol study

CONTACTS AND LOCATIONS:
Overall Officials: M Elhafeez Assistant Professor Obstetrics and Gy, phD, Study Director — Obstetrics and Gynecology; H Fathy Assistant Professor Obstetrics and Gy, phD, Study Director — ASU
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Abbasyia
  - Ain Shams University, Cairo

REFERENCES:
- [Result] Benati M, Montagnana M, Danese E, Paviati E, Giudici S, Ruzzenente O, Franchi M, Lippi G. The clinical significance of DJ-1 and HE4 in patients with endometrial cancer. J Clin Lab Anal. 2018 Jan;32(1):e22223. doi: 10.1002/jcla.22223. Epub 2017 Apr 4. PMID 28374920
- See also: endometrial cancer — http://www.ncbi.nlm.nih.gov/pubmed/28374920